CLINICAL TRIAL: NCT05572840
Title: Wear Your Mask, Wash Your Hands, Don't Get COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Aylin Kurt, Lecturer, Bartın Unıversity
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-SBB-0209
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Coronavirus; Child, Only
MeSH Terms: conditions — Coronavirus Infections | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training and activities (Experimental): The training program consists of two modules. The 1st module consists of a theoretical lecture (PowerPoint presentation) and an activity (application of hygienic handwashing by the researcher) explaining what to do for hygienic handwashing. The 2nd module consists of the theoretical explanation (PowerPoint presentation) in which the correct mask usage is explained and the activity (the "make your own mask" activity by painting the masks).
  Interventions: Other: Training and activities

INTERVENTIONS:
Other: Training and activities — The training program consists of two modules. The 1st module consists of a theoretical lecture (powerpoint presentation) and an activity (application of hygienic handwashing by the researcher) explaining what to do for hygienic handwashing. The 2nd module consists of the theoretical explanation (powerpoint presentation) in which the correct mask usage is explained and the activity (the "make your own mask" activity by painting the masks).

SUMMARY:
The aim of this project is to determine the effect of training given to children aged 11-14 on hand hygiene and mask use. In line with this general purpose, the hypotheses of the research are as follows:

H0= Education given to children aged 11-14 on hand hygiene and mask use has no effect on children's hand hygiene and mask use behaviors.

H1= With the education given to children aged 11-14 on hand hygiene and mask use, children will exhibit more correct hand hygiene and mask use behaviors.

DETAILED DESCRIPTION:
The universe of the research will consist of 273 secondary school students between the ages of 11-14 according to the education and training of Bartın Ertuğrul Gazi Secondary School. The children's inclusion criteria are as follows:

* Being between the ages of 11-14,
* Being a student of Bartın Ertuğrul Gazi Secondary School,
* The child and his parents agree to participate in the project,
* The child's speech and visual impairment do not have any handicap that would force or hinder communication.

Intervention: Once enrolled and consent is documented, eligible subjects will participate in the study for approximately three months. Participants will be expected to attend 2 training sessions and 2 activities (wearing masks and hygienic hand washing), each is up to one hour in length. Follow-up will be made at the beginning of the training, right after the last training. Data analysis will begin once all trainings and activities have been completed. Investigators anticipate completing the study, including primary analyses, within six months from the date recruitment begins.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 11-14,
* Being a student of Bartın Ertuğrul Gazi Secondary School,
* The child and his parents agree to participate in the project,
* The child's speech and visual impairment do not have any handicap that would force or hinder communication.

Exclusion Criteria:

* Not to be between the ages of 11-14,
* Not being a student of Bartın Ertuğrul Gazi Secondary School,
* The child and his parents do not agree to participate in the project,
* The child's speech and vision impairment, or any disability that would force or hinder communication.

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 273 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Change of the mean scores obtained by the children in the intervention group from the "Hand Hygiene Behavior Form" before and after the trainings and activities | 6 months
  "Hand Hygiene Behavior Form" will be completed before the training and activities that gather quantitative data that will address hand hygiene behavior in children. A minimum of 0 points and a maximum of 42 points can be obtained from the form. The higher scores mean the higher proper hand hygien behaviors. This scale will also be completed after the training and activities. The quantitative data will be used to measure the change in the children's hand hygiene behavior before, and after the proposed intervention. Data will be analyzed using Statistical Package for the Social Sciences package program.
Change of the mean scores obtained by the children in the intervention group from the "Behavior Form for Using Masks" before and after the trainings and activities | 6 months
  "Behavior Form for Using Masks" will be completed before the training and activities that gathers quantitative data that will address using masks behavior in children. A minimum of 0 points and a maximum of 42 points can be obtained from the form. The higher scores mean the higher proper using masks behaviors. This scale will also be completed after the training and activities. The quantitative data will be used to measure the change in the children's using masks behavior before, and after the proposed intervention. Data will be analyzed using Statistical Package for the Social Sciences package program.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartin Ertugrul Gazi Secondary School, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol